CLINICAL TRIAL: NCT07069218
Title: Efficacy of Two Hydroxyapatite-Based Toothpastes on Enamel Remineralization: A Randomized Controlled Trial
Brief Title: Hydroxyapatite Toothpastes and Enamel Remineralization:
Acronym: HEREMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-REMINEN
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Enamel Hypomineralization; Tooth Erosion
Keywords: Hydroxyapatite Toothpaste; Enamel Remineralization; DIAGNOcam; DIAGNOdent; Tooth Erosion; Dentin Sensitivity; Dental Plaque; Oral Health; Randomized Controlled Trial; Preventive Dentistry
MeSH Terms: conditions — Dental Enamel Hypomineralization; Tooth Erosion; Dentin Sensitivity; Dental Plaque | interventions — Toothpastes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biorepair Group (Experimental): Participants receive professional oral hygiene sessions every 3 months and use Biorepair® Total Protection Plus toothpaste (biomimetic microRepair-based) twice daily for 6 months.
  Interventions: Drug: Biorepair® Total Protection Plus Toothpaste
- Bioniq Group (Active Comparator): Participants receive professional oral hygiene sessions every 3 months and use Bioniq® Repair toothpaste (conventional hydroxyapatite-based) twice daily for 6 months.
  Interventions: Drug: Bioniq® Toothpaste

INTERVENTIONS:
Drug: Biorepair® Total Protection Plus Toothpaste — Participants will use Biorepair® Total Protection Plus toothpaste twice daily for 6 months. The toothpaste contains biomimetic microRepair® particles based on zinc-substituted hydroxyapatite, intended to promote enamel remineralization, reduce sensitivity, and protect against erosion and plaque accumulation. Professional dental cleanings will also be performed every 3 months.
  Arms: Biorepair Group
Drug: Bioniq® Toothpaste — Participants will use Bioniq® Repair toothpaste twice daily for 6 months. The toothpaste contains 20% conventional hydroxyapatite and is designed to restore enamel, reduce dentin hypersensitivity, and protect against erosion. Professional dental cleanings will also be performed every 3 months.
  Arms: Bioniq Group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the efficacy of two commercially available toothpastes containing hydroxyapatite in the remineralization of early enamel lesions. The study compares Biorepair® Total Protection Plus, which contains biomimetic microRepair particles, with Bioniq® Repair, a conventional hydroxyapatite-based toothpaste.

Forty participants will be randomly assigned to either the trial group (Biorepair®) or the control group (Bioniq®), and both groups will receive quarterly professional dental cleanings and use the assigned toothpaste twice daily for 6 months.

The primary outcome is the change in enamel demineralization, assessed by DIAGNOdent Pen scores, in permanent molar fissures and upper central incisors. Secondary outcomes include enamel integrity assessed by DIAGNOcam imaging and ICDAS scores, as well as changes in dental sensitivity (Schiff Air Index), erosive wear (BEWE Index), plaque accumulation (Plaque Index), gingival inflammation (Bleeding Index), and extrinsic stains (Modified Lobene Stain Index). Patient satisfaction will also be evaluated at the end of the study using a self-administered questionnaire.

This study will help determine whether biomimetic hydroxyapatite offers superior benefits in maintaining enamel health compared to conventional formulations, supporting evidence-based preventive strategies in dental care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 6 and 18 years
* Ability to understand and follow instructions in Italian or English
* Signed written informed consent provided by the parent/legal guardian and assent from the minor
* Good cooperation and adherence to clinical instructions
* Fully erupted permanent first molars and upper central incisors in good general condition
* DIAGNOdent Pen baseline values in the C1 (0-12) or C2 (13-24) range

Exclusion Criteria:

* DIAGNOdent Pen values greater than 25
* Ongoing systemic antibiotic therapy
* Presence of sealants or composite restorations on first permanent molars or upper central incisors
* Severe enamel alterations such as molar-incisor hypomineralization (MIH), fluorosis, or extensive white/brown spot lesions
* Poor motivation or limited compliance with study procedures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in DIAGNOdent Pen values in enamel fissures and upper central incisors | Baseline to 6 months (T0-T3)
  o assess the remineralizing efficacy of biomimetic hydroxyapatite (Biorepair® Total Protection Plus) compared to conventional hydroxyapatite (Bioniq® Repair) by evaluating the reduction in DIAGNOdent Pen fluorescence values recorded in the occlusal fissures of permanent molars and on the surfaces of upper central incisors. Measurements will be taken at four timepoints (T0, T1, T2, T3) over a 6-month period.
  The DIAGNOdent Pen provides a numerical score (0-99) based on laser fluorescence, where higher values indicate increased enamel demineralization. Lower values after treatment reflect improved enamel health and remineralization.

SECONDARY OUTCOMES:
Change in ICDAS Scores via DIAGNOcam Imaging | Baseline to 6 months (T0-T3)
  To assess enamel demineralization using the International Caries Detection and Assessment System (ICDAS) recorded through DIAGNOcam transillumination images. The PI will assign ICDAS scores to the occlusal surfaces of permanent molars and labial surfaces of upper central incisors at each timepoint. The ICDAS scoring system ranges from 0 to 6, where a score of 0 indicates sound tooth structure, scores of 1 and 2 represent initial changes in enamel, and scores from 3 to 6 reflect progressive levels of localized enamel breakdown and cavitation. A decrease in score over time is interpreted as a sign of remineralization or lesion arrest.
Change in Dentin Hypersensitivity Using Schiff Air Index | Baseline to 6 months (T0-T3)
  To evaluate dentin hypersensitivity in response to an air stimulus applied to exposed cervical surfaces using the Schiff Air Index. The clinician will assign a score from 0 to 3, where a score of 0 indicates no reaction, 1 indicates a reaction without the patient requesting discontinuation, 2 indicates a reaction and a request to stop, and 3 indicates a strong reaction and immediate request to discontinue. The score reflects the participant's response to air-blast stimulation and will be recorded at each timepoint. A decrease in score suggests reduced hypersensitivity.
Change in Enamel Erosion Using BEWE Index | Baseline to 6 months (T0-T3)
  To monitor changes in enamel erosion using the Basic Erosive Wear Examination (BEWE) index. The examiner will assess each sextant and assign a score from 0 to 3. A score of 0 indicates no erosive tooth wear, a score of 1 indicates initial surface loss, a score of 2 represents distinct defects with hard tissue loss involving less than 50% of the surface area, and a score of 3 indicates hard tissue loss affecting more than 50% of the surface. The highest score per sextant is recorded, and a cumulative BEWE score is calculated for each participant at every timepoint. A reduction in the BEWE score suggests improved enamel preservation.
Change in Plaque Accumulation Using Plaque Index | Baseline to 6 months (T0-T3)
  To evaluate changes in plaque accumulation between groups using the Plaque Index (Silness and Löe, 1964), which measures plaque thickness along the gingival margin. The scoring system ranges from 0 to 3. A score of 0 indicates no plaque. A score of 1 corresponds to a thin film of plaque adhering to the free gingival margin and adjacent area of the tooth, which is only detectable by running a probe across the tooth surface. A score of 2 represents moderate accumulation of soft deposits visible to the naked eye, either on the tooth surface or within the gingival margin. A score of 3 indicates heavy accumulation of soft debris in the gingival pocket or on the tooth and gingival margin. The PI assigns a score for each examined surface, and the average value per participant is calculated at each timepoint (T0-T3).
Change in Gingival Inflammation Using Bleeding Index | Baseline to 6 months (T0-T3)
  To assess changes in gingival inflammation by comparing Bleeding Index (BI) values between groups at each study timepoint. The clinician will gently probe the gingival sulcus of selected teeth and assign a score from 0 to 3 for each site. A score of 0 indicates no bleeding after probing. A score of 1 indicates isolated bleeding spots visible after probing. A score of 2 indicates a line of blood along the gingival margin. A score of 3 indicates profuse bleeding immediately after probing. The average score per participant will be calculated based on all examined sites at each timepoint. Higher scores reflect greater gingival inflammation.
Change in Extrinsic Staining Using Modified Lobene Stain Index | Baseline to 6 months (T0-T3)
  To evaluate changes in extrinsic dental staining using the Modified Lobene Stain Index, which assesses both the area and intensity of stain on selected tooth surfaces. The PI assigns a score from 0 to 3 for the area of stain, where 0 indicates no staining and 3 indicates stain covering more than two-thirds of the surface. Separately, the intensity of stain is scored from 0 to 3, where 0 indicates no stain and 3 indicates heavy dark staining. The final index is obtained by multiplying the area score by the intensity score. Higher values reflect more extensive and intense staining. Measurements are collected at baseline and at each follow-up (T0-T3).
Patient Satisfaction via Self-Administered Questionnaire | At 6 months (T3 only)
  To evaluate subjective satisfaction with the assigned toothpaste at the end of the study using a self-administered questionnaire. Participants will rate various aspects such as taste, texture, perceived effectiveness, and overall satisfaction. The PI will collect and score responses using a standardized Likert-type scale ranging from 1 (very dissatisfied) to 5 (very satisfied). The mean satisfaction score per participant will be analyzed and compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.